CLINICAL TRIAL: NCT02423980
Title: G-Pen™ (Glucagon Injection) for Induced Hypoglycemia Rescue in Adult Patients With T1D
Brief Title: G-Pen™ for Hypoglycemia Rescue in T1D Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XSGP-202
Record Dates: First submitted 2015-04-09; First posted 2015-04-22 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucagon (Experimental): 1 mg G-Pen™ (glucagon injection) first, followed by 0.5 mg
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon
  Other Names: G-Pen™ (glucagon injection)

SUMMARY:
This is an open-label, exploratory pilot study in patients with T1D. The study will involve two daytime clinical research center visits 7-14 days apart. Subjects will receive a single injection of G-Pen™ (glucagon injection) at each visit.

DETAILED DESCRIPTION:
Following eligibility confirmation, each study participant will undergo two episodes of insulin-induced hypoglycemia with plasma glucose < 50 mg/dL. Both episodes will be treated with a single subcutaneous injection of G-Pen™ glucagon. For the first treatment visit, all subjects will receive a 1 mg dose of G-Pen™ glucagon. The investigator will have discretion to repeat this same dose at the second treatment visit or give a 0.5 mg dose of G-Pen™ glucagon. A follow-up phone call will be conducted 3-7 days following administration of the final dose of study drug as a safety check.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 24 months

Exclusion Criteria:

* Pregnant or Lactating
* HbA1c >10.5% at screening
* Use of > 2.0 U/kg total insulin dose per day
* Inadequate bilateral venous access in both arms
* Renal insufficiency
* Congestive heart failure, NYHA class II, III or IV
* Active malignancy within 5 years from screening
* Major surgical operation within 30 days prior to screening
* Seizure or bleeding disorder
* Glycogen storage disease
* Active substance or alchohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diablo Clinical Research, Inc., Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 adults with type 1 diabetes were recruited at a clinical research center over a period of 1 month.
Pre-assignment Details: One subject was given the 1 mg dose of glucagon at both treatment visits, so only 6 subjects received the 0.5 mg dose.
Groups:
- G-Pen™ (Glucagon Injection) 1 mg First, Followed by 0.5 mg: A 1 mg dose of glucagon at an initial clinic visit, followed by a 0.5 mg dose of glucagon given at a subsequent clinic visit after a 1-2 week wash-out.
Period: Overall Study
Arm/Group | G-Pen™ (Glucagon Injection) 1 mg First, Followed by 0.5 mg
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- G-Pen™ (Glucagon Injection) 1 mg First, Followed by 0.5 mg: A 1 mg dose of G-Pen was given at an initial clinic visit. After a 1-2 week wash-out, subjects received a 0.5 mg dose of G-Pen™ at a second visit.
Arm/Group | G-Pen™ (Glucagon Injection) 1 mg First, Followed by 0.5 mg
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 42 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasma Glucose > 70 mg/dL at 30 Minutes Post-treatment
Description: For 90 minutes following treatment, plasma glucose was measured every 5 minutes, with an increase in plasma glucose to >70 mg/dL within 30 minutes of treatment being considered a positive response.
Time Frame: 0-90 minutes
Population: All treated subjects
Measure: Number; unit: participants with positive response
Groups:
- Glucagon 1 mg: 1 mg G-Pen™ (glucagon injection)
  Glucagon
- Glucagon 0.5 mg: 0.5 mg G-Pen™ (glucagon injection)
  Glucagon
Arm/Group | Glucagon 1 mg | Glucagon 0.5 mg
Number analyzed (Participants) | 7 | 6
participants with positive response | 7 | 6

2. Secondary Outcome: Time to Plasma Glucose > 70 mg/dL
Description: Following treatment, plasma glucose was measured every 5 minutes. The first such measurement at which plasma glucose concentration was observed to be >70 mg/dL was reported as the time to response.
Time Frame: 0-90 minutes
Population: All treated subjects
Measure: Median (Full Range); unit: minutes
Arm/Group | Glucagon 1 mg | Glucagon 0.5 mg
Number analyzed (Participants) | 7 | 6
minutes | 15 [10 to 20] | 15 [10 to 20]

3. Secondary Outcome: Time to Resolution of Induced Hypoglycemia Symptoms
Description: Prior to and every 5 minutes after treatment, subjects were asked to rate the severity of each of 8 symptoms on a scale from 1 to 6, with 1 indicating the symptom was absent and 6 indicating the symptom was severe. The sum of the scores for the 8 individual symptoms was reported as the total hypoglycemia symptom score, which ranged from 8-48. The first time point post-treatment at which total hypoglycemia symptom score = 8 (i.e., all symptoms were absent) was considered the time to resolution. One and two subjects were unevaluable for response to the 1 mg and 0.5 mg doses of glucagon, respectively, as they reported no symptoms (i.e., total symptom score = 8) prior to treatment.
Time Frame: 0-30 minutes
Population: Subjects with symptoms of hypoglycemia at time of treatment
Measure: Median (Full Range); unit: minutes
Arm/Group | Glucagon 1 mg | Glucagon 0.5 mg
Number analyzed (Participants) | 6 | 4
minutes | 20 [5 to 30] | 27.5 [25 to 30]

ADVERSE EVENTS:
Time Frame: Total evaluation time was up to 3 weeks per subject.
Description: Treatment-emergent events observed during the dosing visits or subsequently reported by the subjects between visits or at the follow-up phone call occurring 3-7 days after the second treatment visit were recorded.
Arm/Group | Glucagon 1 mg | Glucagon 0.5 mg
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/7 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon 1 mg (N=7) | Glucagon 0.5 mg (N=6)
Vasovagal syncope (Nervous system disorders) | 1 (1) | 0 (0) — While consuming the post-study meal at approximately 90 minutes post-dosing, subject became nauseated and subsequently vomited and fainted.Subject recovered with no sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon 1 mg (N=7) | Glucagon 0.5 mg (N=6)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No